CLINICAL TRIAL: NCT05948306
Title: The Effects of Patient-Centred Skin Care on Barrier Functions of Skin in Critical Patients: Randomised-Controlled Trial
Brief Title: Effects of Patient-centered Skin Care in Critical Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Bilgi University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other); University of Southampton (Other)
Responsible Party: Principal Investigator, TUĞBA YENİ, Lecturer, Koç University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022/81
Record Dates: First submitted 2023-03-27; First posted 2023-07-17 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Pressure Injury; Transepidermal Water Loss; sk
Keywords: pressure injury; patient-centered care; skin care protocol; transepidermal waterloss; skin properties
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: This study was planned as a randomized controlled trial including experimental and control groups.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient-centered skin care group (Experimental): A patient-centered skin care protocol developed according to the Stetler Model will be applied to the experimental group.
  Interventions: Other: Critical Patient-Centered Skin Care Protocol
- Routine skin care group (No Intervention): The routine skin care of the ICU will be applied to the control group during the study.

INTERVENTIONS:
Other: Critical Patient-Centered Skin Care Protocol — A patient-centered skin care protocol prepared by the researchers in accordance with the Stetler Model will be applied to the experimental group.
  Sub-titles of this protocol; evaluation of risk factors, examination of the skin from head to toe, skin hygiene, examining the effects of critical illness on the skin, mobilization and re-positioning, incontinence management, maintaining nutrition, and using a support surface. For each sub-heading, application items regarding patient demands and suggestions will be added.
  Arms: Patient-centered skin care group

SUMMARY:
Many critical diseases can damage skin and tissue integrity due to natural immobility, hemodynamic instability, poor tissue perfusion, use of medical devices and many other internal and external factors. Skin damage frequently seen in intensive care units; It can be listed as skin tears and secondary cutaneous infections, especially pressure injuries (PI) and incontinence-associated dermatitis (IAD). In the DecubICU's study, which has the largest sample number ever, published in 2021, the prevalence of pressure ulcers and related factors in 1117 intensive care units from 90 different countries were evaluated; Pressure ulcers were detected in 6747 of 13,254 patients hospitalized in the ICU, and 57% of these wounds were reported to be associated with the intensive care unit.

In addition to pressure injuries, another skin problem that has also been focused on in nursing science in the last 10 years; incontinence-associated dermatitis. IAD, which develops on the skin exposed to urine and faeces, is not only a skin damage that needs to be examined on its own, but also paves the way for the development of pressure sores and can also progress together with pressure injuries. The study which was published in 2018, examined 109 intensive care patients, while the incidence of IAD was determined as 23.6%, while in 2019 another study in which 351 patients were included for 52 weeks, annual prevalence of IAD ranged from 17% and weekly incidences ranged from 0-70%. The findings of three different studies conducted in the intensive care unit are that IAD developed in 6% of 112 patients, 26.2% of 145 patients, and 65.4% of 266 patients, respectively. However, despite the limited literature, the high prevalence rates and the strong relationship between pressure injuries and incontinence associated dermatitis point to the necessity of evaluating these two skin injuries together.

Each existing skin injury reduces the quality of life by causing pain and pain to the individual, and also increases hospitalizations and infection rates, placing a financial burden on the health system and causing loss of workforce. For all these reasons, skin problems are considered as a quality indicator in hospitals and the primary responsibility for maintaining skin integrity is attributed to nurses. Guidelines published by EPUAP, National Pressure Injury Advisory Panel and Pan Pacific Pressure Injury Alliance (PPPIA) in 2019 in the prevention of pressure injuries in intensive care units play a key role in determining nurses' attempts to preserve skin and tissue integrity. In the prevention of incontinence-related dermatitis, the best practices guide published by Dimitri Beckmann in 2015 should be integrated into clinics.

Furthermore, the person-centered approach in skin care has been considered as a concept that should be focused on by the authors in recent years, and in a systematic review published in 2020, clinical applications of the person-centered care approach in wound care were suggested by considering the current evidence. However, the resources in which prevention strategies are focused on individual-centered care are very limited. Therefore, in this study, it was aimed to develop a critical patient-centered skin care protocol and to examine the effects of this protocol on the barrier functions of the skin.

HYPOTHESES AND DETAILED AIMS ARE BELOW.

The primary aim of the study is to examine the effect of critical patient centered skin care on the barrier function of the skin. The hypotheses for the primary purpose of this study are as follows:

* H1a: The mean TEWL is lower in ICU patients receiving patient-centred care than in those receiving standard care.
* H1b: The mean skin pH is more acidic in ICU patients receiving patient-centred care than in those receiving standard care.
* H1c: The PI risk is lower in ICU patients receiving patient-centred care than in those receiving standard care.
* H1d: The incidence of PI is lower in ICU patients receiving patient-centred care than in those receiving standard care.

ELIGIBILITY:
Inclusion Criteria:

* Taking care in the ICU for 24 hours as a stable patient,
* Glasgow coma scale to be at least 10 points,
* Having at least one of the urinary/fecal/mixed incontinence types,
* Being treated in the intensive care unit for at least 7 days,
* Being over 18 years old

Exclusion Criteria:

* Being after cardiopulmonary resuscitation (post CPR),
* Brain death has occurred,
* Having had multiple trauma,
* Being diagnosed with allergic asthma
* Having any skin health problem before ICU admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2023-09-27 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-12 (Actual)

PRIMARY OUTCOMES:
Change of transepidermal water loss | This parameter will be measured through study completion for every day
  This outcome includes transepidermal water loss. It will be assessed by researcher with VapoMeter.
Change of skin pH | This parameter will be measured through study completion for every day
  This outcome includes skin pH changing. It will be assessed by researcher with pHmeter.

SECONDARY OUTCOMES:
Incidence of pressure injuries | Patients included during the study will be followed for at least 4 days or through the hospitalization
  Pressure injuries will be assessed according to the EPUAP stage system
Risk score of pressure injuries | Patients included during the study will be followed for at least 4 days or through the hospitalization
  Scale is used for risk detection

CONTACTS AND LOCATIONS:
Locations (1):
- Beykoz State Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All results of the project will be shared by researcher via publishing.
Supporting Information: Study Protocol, CSR
Time Frame: Sharing will be possible in a year. And it is available for unlimited time. Tugba Yeni as a first author is responsible for sharing.
Access Criteria: Researcher worked with ICU patients and tissue viability can access to research results.

REFERENCES:
- [Result] Campbell J, Cook JL, Doubrovsky A, Vann A, McNamara G, Coyer F. Exploring Incontinence-Associated Dermatitis in a Single Center Intensive Care Unit: A Longitudinal Point Prevalence Survey. J Wound Ostomy Continence Nurs. 2019 Sep/Oct;46(5):401-407. doi: 10.1097/WON.0000000000000571. PMID 31513128
- [Result] Gethin G, Probst S, Stryja J, Christiansen N, Price P. Evidence for person-centred care in chronic wound care: A systematic review and recommendations for practice. J Wound Care. 2020 Sep 1;29(Sup9b):S1-S22. doi: 10.12968/jowc.2020.29.Sup9b.S1. PMID 32935648
- [Result] Johansen E, Lind R, Sjobo B, Petosic A. Moisture associated skin damage (MASD) in intensive care patients: A Norwegian point-prevalence study. Intensive Crit Care Nurs. 2020 Oct;60:102889. doi: 10.1016/j.iccn.2020.102889. Epub 2020 Jun 11. PMID 32536519
- [Result] Telser E. [Pharmaceutic incompatibilities--pharmaceutically undesirable conditions--in feed drugs. II. Chemical incompatibilities]. Dtsch Tierarztl Wochenschr. 1979 Feb 5;86(2):69-73. No abstract available. German. PMID 33034
- [Result] Valls-Matarin J, Del Cotillo-Fuente M, Ribal-Prior R, Pujol-Vila M, Sandalinas-Mulero I. Incidence of moisture-associated skin damage in an intensive care unit. Enferm Intensiva. 2017 Jan-Mar;28(1):13-20. doi: 10.1016/j.enfi.2016.11.001. Epub 2017 Jan 16. English, Spanish. PMID 28110903
- [Result] Wang X, Zhang Y, Zhang X, Zhao X, Xian H. Incidence and risk factors of incontinence-associated dermatitis among patients in the intensive care unit. J Clin Nurs. 2018 Nov;27(21-22):4150-4157. doi: 10.1111/jocn.14594. Epub 2018 Jul 26. PMID 29964368
- [Result] Wei L, Bao Y, Chai Q, Zheng J, Xu W. Determining Risk Factors to Develop a Predictive Model of Incontinence-associated Dermatitis Among Critically Ill Patients with Fecal Incontinence: A Prospective, Quantitative Study. Wound Manag Prev. 2019 Apr;65(4):24-33. PMID 30994472
- [Result] European Pressure Ulcer Advisory Panel, National Pressure Injury Advisory Panel and Pan Pacific Pressure Injury Alliance. Prevention and Treatment of Pressure Ulcers/Injuries: Quick Reference Guide. Emily Haesler (Ed.). EPUAP/NPIAP/PPPIA: 2019.
- [Result] Beeckman D et al. Proceedings of the Global IAD Expert Panel. Incontinence- associated dermatitis: moving prevention forward. Wounds International 2015.